CLINICAL TRIAL: NCT02833116
Title: Efficacy and Safety of Dexamethasone Versus Betamethasone Epidural Caudal Administration for Treatment of Lumbosacral Radiculalgia: Randomized Clinical Trial
Brief Title: Epidural Dexamethasone Versus Betamethasone for Treatment of Lumbosacral Radiculalgia
Acronym: BetaDexaCaudal
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Enrique Manuel Barez Hernandez, Medical Doctor, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Beta-Dexa-Caudal
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Pain
Keywords: radiculalgia; chronic pain; quality of life
MeSH Terms: conditions — Chronic Pain | interventions — Betamethasone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Betamethasone (Experimental): One ampule containing 12 mg of betamethasone in a syringe of 10 ml
  Interventions: Drug: Betamethasone
- Group Dexamethasone (Active Comparator): One ampule containing 4 mg of dexamethasone in a syringe os 10 ml
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Betamethasone
  Arms: Group Betamethasone
Drug: Dexamethasone
  Arms: Group Dexamethasone

SUMMARY:
This study evaluate the administration of epidural betamethasone versus dexamethasone for pain reduction, consumption of analgesic and quality of life. Half of the patient will receive dexametasone and the other half betametasone.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral leg pain secondary to lateral stenosis, disc protrusion or herniated disc.
* Age between 18 and 80 years.
* Moderate to severe pain (NVS>4).
* Right proficient oral and written language.

Exclusion Criteria:

* Patients with high intracranial pressure.
* Patients with Multiple Sclerosis.
* Patients with Guillain-Barré syndrome radiculopathy of vascular origin.
* Patients with previous lumbar surgery.
* Patients pregnant or lactating.
* Patients with allergy or intolerance to any of the drugs used.
* Patients with severe cognitive impairment.
* Patients with intrathecal injectio radiculalgia.
* Patients with poorly controlled major psychiatric pathology.
* Patients with type I diabetes or poorly controlled type II diabetes (Hb1Ac>8.5).
* Patients with glaucoma.
* Patients with caudal equine syndrome.
* Patients with pre-treatment with steroid injections/or local anesthetics.
* Patients with central canal stenosis.
* patients with chronic treatment with oral corticosteroids without stabilized pattern.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Pain. | 3 months.
  Pain according to numerical visual pain scale.

SECONDARY OUTCOMES:
Quality of life. | 7 days, 1, 3 and 6 months.
  Quality of life according to SF-36.
Pain. | 7 days, 1, 3 and 6 months.
  Pain according to numerical visual pain scale.
Adverse events. | 7 days, 1, 3 and 6 months.
  Adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Barez, Principal Investigator — Basque Health Service: Araba University Hospital; Borja Mugabure, Study Director — Basque Health Service: Donosti University Hospital; Fernando Torre, Principal Investigator — Basque Health Service: Galdakao University Hospital
Locations (1):
- Enrique Barez, Vitoria-Gasteiz, Álava, Spain

IPD SHARING:
Plan to Share IPD: No